CLINICAL TRIAL: NCT03262805
Title: To Assess the Lanconone® (E-OA-07) Efficacy in Physical Activity-related Pain- LEAP Study
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EB/170401/LC/OA
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee OA; Joint Pain; Dietary supplement; WOMAC; Lequesne index; hs-CRP
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Active (Active Comparator): Lanconone(R)
  Interventions: Dietary Supplement: Lanconone

INTERVENTIONS:
Dietary Supplement: Lanconone — . Lanconone® is a joint pain supplement containing natural herbs such as Shyonak, Ashwagandha, Shunthi, Guggul, Chopchini, Rasna and Shallaki in therapeutic quantities and documented in the ancient scriptures as pain relievers.
  Arms: Active
Other: Placebo — Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The current study is designed to assess the pain relieving effect of 4-weeks ingestion of this commercialized dietary supplement (Lanconone®, Enovate Biolife, LLC, 1000 mg twice per day) in mild to moderate OA subjects. Also, the current study intends to assess the safety and efficacy of long term administration of Lanconone in larger sample size as compared to the earlier studies.15,16 The study also intends to analyse the effect on joint stiffness and function by means of self-reported WOMAC & Lequesne questionnaire.The effect of IP on clinically proven biomarker, hs-CRP will be analyzed in comparison with placebo.

DETAILED DESCRIPTION:
This study has been planned to evaluate the efficacy of Lanconone® in enhancing the overall joint health in the population of ≥ 40 years of age during the daily life activities by the reduction of the joint pain and discomfort. Assessment of pain is the primary objective which will be done by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the severity of osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The early onset of action (3 days after commencement of the IP administration) for pain relief which was not captured in the past studies, will be captured in the current study by the telephonic assessment of the study subjects. Lequesne et al developed an index of severity for osteoarthritis for the knee which can be used to assess the effectiveness of therapeutic interventions. Unlike the earlier studies, we will use the Lequesne Functional Index (LFI) to assess the extent of joint health degeneration. In relation to OA, elevated levels of hs-CRP have been correlated with symptoms of joint pain and stiffness. Hence, we decided to analyze the hs-crp levels as one of the secondary objectives. Also, the rescue medication consumption has been limited to lower per day consumption compared to earlier studies to avoid the placebo effect influence on the study results. The efficacy of the IP in sustaining the pain relieving effect will be analyzed on day 35, i.e. one week after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* M/F subject aged ≥ 40 to ≤ 65 with unilateral or bilateral OA of the knee for greater than 3 months as presented by pain in knee.
* Body mass index (BMI) must be 25 to 29.9 kg/m2.
* WOMAC pain score for index joint: 10 to 16.
* Physically active subjects as indicated by day to day involvement in the mentioned physical activity namely:
* Daily walk of 500 to 1000 meters.
* Routine activities such as descending/ ascending stairs, standing up from a chair; bending to floor; travelling by public transport, domestic cleaning etc.
* Climbing 1 or more fleets of stairs.
* Osteoarthritis grade I/ II (Kellgren-Lawrence classification) as confirmed by radiographic evidence.

Exclusion Criteria:

* Subjects with a history of any joint replacement surgery.
* Subjects not willing to abstain from use of NSAIDs (including low dose aspirin 50 mg/day for cardiovascular health) or herbal/ nutraceutical supplements for joint health/ local analgesics or other traditional pain relieving therapies such as message or acupuncture etc. during the study duration will be excluded.
* Subject with uncontrolled hypertension (blood pressure: systolic ≥140 mm Hg or diastolic ≥ 100 mm Hg) at screening.
* Subjects with history of thyroid hormone derangement will have to provide a recent (within 3 months) thyroid profile report indicative of euthyroid status.
* Use of any immunosuppressive drugs in the last 12 months.
* Use of any corticosteroids drugs in the last 3 months.
* Subject unwilling to refrain from analgesic measures at least 48 hours before each site visit.
* FBS >140 mg/dl.
* History of restless leg syndrome.
* Glucocorticoid injection or hyaluronic acid injection in affected joint within 3 months prior to enrolment.
* Subjects with a chronic pain syndrome and in the judgment of the Investigator is unlikely to respond to any therapy.
* Smokers and tobacco users.
* Alcohol consumption of more than 200 ml/ week
* History of surgery in lower limb.
* Subjects suffering from diabetic neuropathy.
* Subjects suffering from deep vein thrombosis.
* Pregnant / lactating women and women who are planning to get pregnant.
* Recent (< 3 months) participation in a clinical study.
* History of major chronic hepatic, cardiovascular, neurological or immunosuppressive conditions or the presence of any infections.
* Subjects with localized trauma to the lower limb.
* A psychiatric condition, chronic alcohol or drug abuse problem as evidenced by withdrawal symptoms.
* Subjects planning to travel in the next 35 days or engage in any non-routine activity that is likely to strain the knees.
* Subject a history of malignancy, active gastrointestinal disease, chronic or acute renal/hepatic disorders, or significant coagulation disorders.
* Subjects on vitamins, nutritional supplement or herbal product since last 2 weeks.
* Subjects otherwise judged by the investigator to be inappropriate for inclusion in the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
WOMAC pain score. | 28 days
  • Change in terms of percentage reduction of joint pain from baseline to Day 28 during daily life activities assessed by WOMAC pain score.

SECONDARY OUTCOMES:
WOMAC stiffness score | 28 days
  Change in terms of percentage reduction of joint pain from baseline to Day 28 joint stiffness as assessed by WOMAC stiffness score.
WOMAC physical performance score. | 28 days
  Change in terms of percentage reduction of joint pain from baseline to Day 28 in physical performance during daily life activities as assessed by WOMAC physical performance score.
Lequesne Functional Index | 28 days
  % reduction in joint degradation process as from baseline to Day 28 as assessed by Lequesne Functional Index
Serum hs-CRP levels. | 28 days
  % reduction in joint pain marker from baseline to Day 28 as assessed by serum hs-CRP levels.
BMI | 28 days
  % change in joint degradation related risk factor from baseline to Day 28 as assessed by BMI.
% responders | 28 days
  Comparison of uniformity of positive pain relieving individual response as assessed by % responders with ≥ 17% reduction in WOMAC pain score at Day 28.
Rescue medication consumption | 28 days
  Comparison of alternate analgesic therapy requirement as assessed by number of rescue medication consumption during the study.
Sustained effect | 35 days
  • To assess the sustained drug free period as assessed by WOMAC pain score joint pain at Day 35 as compared to Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastava, MD, Study Director — Enovate Biolife Pvt Ltd
Locations (3):
- India (3):
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Kewalramani's Clinic, Mumbai, Maharashtra
  - KK Medical Centre, Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Girandola RN, Srivastava S, Loullis CC. A clinical trial comparing Lanconone(R) with ibuprofen for rapid relief in acute joint pain. Trials. 2016 Apr 6;17:189. doi: 10.1186/s13063-016-1268-6. PMID 27052991